CLINICAL TRIAL: NCT06351969
Title: Evaluating Placental Thickness and Thickness of Uterine Muscle at Placenta Attachment in Prediction of Postpartum Blood Loss in Placenta Accreta
Status: Not yet recruiting | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelsalam Ahmed Abdelhamid, Principal Investigator, Benha University
Other Study IDs: 1111
Record Dates: First submitted 2024-03-28; First posted 2024-04-08 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Post Partum Hemorrhage
Keywords: Post Partum Hemorrhage; placental thickness; cesarean section; vaginal delivery
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aim of the Work is To determine the significance of the placental thickness and the thickness of the uterine muscle layer at placental attachment in the prediction of postpartum hemorrhage in cases of placenta previa accreta and to evaluate both of them as as parameters for identifying high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy (37 wk gastation and more )
* Single viable fetus

Exclusion Criteria:

* Severe hematological disorders that could cause abnormal coagulation
* Previous history of PPH
* twins
* Preterm labour
* IUFD

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: The study will be carried out on 100 pregnant women, who will undergo delivery either by vaginal delivery or cesarean section either as elective palnned at operative list or admitted to Obstetrics ER after complete clinical evaluation
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluating Placental Thickness in cm and Thickness of Uterine Muscle in cm at Placenta Attachment in Prediction of Postpartum Blood Loss in placenta accreta | follow up blood loss in ml intraoperative and 24 hour post operative
  Evaluating Placental Thickness and Thickness of Uterine Muscle at Placenta Attachment in Prediction of Postpartum Blood Loss in placenta accreta

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Benha University, Banhā, benha
  - B Univeristy, Banī Suwayf

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WOMAN Trial Collaborators. Effect of early tranexamic acid administration on mortality, hysterectomy, and other morbidities in women with post-partum haemorrhage (WOMAN): an international, randomised, double-blind, placebo-controlled trial. Lancet. 2017 May 27;389(10084):2105-2116. doi: 10.1016/S0140-6736(17)30638-4. Epub 2017 Apr 26. PMID 28456509
- [Background] Widmer M, Piaggio G, Nguyen TMH, Osoti A, Owa OO, Misra S, Coomarasamy A, Abdel-Aleem H, Mallapur AA, Qureshi Z, Lumbiganon P, Patel AB, Carroli G, Fawole B, Goudar SS, Pujar YV, Neilson J, Hofmeyr GJ, Su LL, Ferreira de Carvalho J, Pandey U, Mugerwa K, Shiragur SS, Byamugisha J, Giordano D, Gulmezoglu AM; WHO CHAMPION Trial Group. Heat-Stable Carbetocin versus Oxytocin to Prevent Hemorrhage after Vaginal Birth. N Engl J Med. 2018 Aug 23;379(8):743-752. doi: 10.1056/NEJMoa1805489. Epub 2018 Jun 27. PMID 29949473
- [Background] Ononge S, Mirembe F, Wandabwa J, Campbell OM. Incidence and risk factors for postpartum hemorrhage in Uganda. Reprod Health. 2016 Apr 14;13:38. doi: 10.1186/s12978-016-0154-8. PMID 27080710
- [Background] Weeks A. The prevention and treatment of postpartum haemorrhage: what do we know, and where do we go to next? BJOG. 2015 Jan;122(2):202-10. doi: 10.1111/1471-0528.13098. Epub 2014 Oct 7. PMID 25289730
- [Background] Liao JB, Buhimschi CS, Norwitz ER. Normal labor: mechanism and duration. Obstet Gynecol Clin North Am. 2005 Jun;32(2):145-64, vii. doi: 10.1016/j.ogc.2005.01.001. PMID 15899352
- [Background] B-Lynch, C., Keith, L., Lalonde, A. & Karoshi, M. (2006). A textbook of postpartum haemorrhage: a comprehensive guide to evaluation,managementand surgical intervention, New Delhi, India, Japee Brothers